CLINICAL TRIAL: NCT02324023
Title: Endoscopic Ultrasound Scanning and Contrast Enhancement for Staging and Evaluation of Angiogenesis of Left Sided Colon Cancers
Brief Title: Endoscopic Ultrasound and Contrast Enhancement for Staging and Evaluation of Angiogenesis of Left Sided Colon Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-4-2014-075
Record Dates: First submitted 2014-11-24; First posted 2014-12-24 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Colonic Neoplasms
Keywords: ultrasound; perfusion; endoscopic
MeSH Terms: conditions — Colonic Neoplasms | interventions — Endosonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic ultrasound and pathology (Experimental): Endoscopic ultrasound and contrast enhanced endoscopic ultrasound for staging and perfusion (preoperatively) compared to pathological stage and vessel density in the pathological specimen (postoperatively).
  Interventions: Device: Endoscopic ultrasound

INTERVENTIONS:
Device: Endoscopic ultrasound — All patients will be evaluated by EUS and CE-EUS, using radial EUS instruments. The EUS scope will be inserted under direct vision, passed by the tumour and examination should begin during withdrawal at 7.5 MHz. The tumour will be characterized describing its echogenicity, echo structure, size, extent into the bowel wall and surrounding structures, and it will be staged using the modification of the TNM classification, based on a five-layer intestinal wall model. The presence/absence of power Doppler signals will be noted. For CE-EUS parameters for objective measurement of tumour perfusion will include maximum intensity of enhancement, mean transit time, time to peak (wash-in time), wash-in slope, area under the curve, representing indirectly blood flow or blood volume in CRC patients.
  Other Names: Endoscopic ultrasonography

SUMMARY:
Cancer in the colon and rectum represents a global health burden being the most common cancer of the digestive tract. It is the second most common cancer in Denmark and only about half of the patients survive this diagnosis. Thorough characterization of the tumour preoperatively is very important, since it determines if the patient should be treated with chemotherapy before operation and, in the future, which operation would be most suitable for the patient.

Research has shown that endoscopic ultrasound (EUS) is superior to a CT-scan, in determining the local growth of the tumour in rectal cancer. Today, a CT-scan is the image modality of choice, and is used in all Danish hospitals when it comes to colon cancer. Hopefully, the investigators can apply EUS in colon cancer patients and thereby alter our diagnostic approach, towards a quicker and safer way to determine which treatment the investigators should offer the patient.

With the screening programme for colorectal cancer in Denmark the investigators will find more and more cases of colorectal cancers, especially in the early stages, before symptoms begin. These small tumours put doctors in several dilemmas concerning the strategy of treatment. Even today, the investigators are very reluctant in offering large-scale operations to elderly and fragile patients who have been diagnosed with cancer in the rectum. Instead, local endoscopic operations are performed in selected patients. This approach has not yet been tried in early colonic cancers. However, it might turn out that local, endoscopic surgery will show to be beneficial for patients with colon cancers and maybe even decrease morbidity, mortality and the regenerative period after surgery.

The aim of this PhD-project is to investigate the utility of the EUS-method in characterizing tumours in the colon and in investigating the blood flow in the tumour.

DETAILED DESCRIPTION:
Introduction Background: Colorectal carcinoma represents a global health burden being the most common cancer of the digestive tract. The lifetime risk of developing colorectal carcinoma is 5%, while the overall number of patients currently alive with diagnosed disease in Denmark is estimated to be 30.000 patients. Approximately 70% of cases involve the colon, with the remaining 30% involving the anus and rectum. The mortality rate is intimately related to its high metastatic ability and therefore prognosis strongly depends on the stage at diagnosis.

Angiogenesis: Angiogenesis plays an important role in tumour growth and its metastatic potential and it has been attracting a lot of attention in the past years, due to possible implications in prognosis stratification, as well as in the targeted treatment of advanced colorectal cancer. Most cancers depend firmly on the development of a new capillary network to allow nutrition of newly formed tumour cells. These newly developed blood vessels are usually highly permeable and allow the access of tumour cells in the general circulation, leading to metastatic progression. Current treatment strategies for patients with advanced colorectal cancer include a combined regimen of cytotoxic and biologic therapy targeting angiogenesis. Thus, there is a great interest in finding alternative imaging tests for assessing the efficacy of antiangiogenic agents earlier in the course of therapy, based on functional imaging of tumour vascularity. The benefit that is seen in the survival of patients with advanced disease by treatment with antiangiogenic drugs can maybe translate in a neoadjuvant setting or an adjuvant setting in patients with stage III cancer or high risk stage II cancer.

Staging: Tumour is described by the TNM classification of malignant tumours (TNM).

Accurate preoperative staging of colon and rectum cancer is the main factor determining the treatment modality for patients and can greatly influence the results. Prognostication and determination of T stage of colon tumours by using computed tomography (CT) scans have been widely discussed in the literature. Endoscopic ultrasound (EUS) has been suggested the staging tool of choice for rectal cancer, when comparing to CT, yet colonic cancers remain to be investigated.

With the Danish National Bowel Cancer Screening Programme, increasing numbers of early cancers are revealed. During recent years local treatment in patients with rectal carcinoma in situ T0 or (T1/T2N0M0) cancers has become more and more accepted and has opened new avenues in treatment of old, comorbid or in other ways, vulnerable patients. As a result of the screening programme clinicians will naturally be placed in new dilemmas in terms of treatment choices, radical versus local excision, for early colonic cancers. Important issues on colonic cancer excisions, are the intramural extent of invasion and the presence or absence of lymphnode metastasis.

EUS: Endoscopic ultrasound (EUS) is a method consisting of an ultrasound transducer mounted on the tip of an endoscope. It has evolved to be useful for both imaging and intervention in the colon and rectum. The investigators chose to use the radial-array endoscope with its 360o view in evaluating colonic cancers, often presenting as circumferential lesions. EUS ability to depict the layers of the GI wall has proven the method usefull in staging GI cancers . Imaging of the blood flow in the vessels and evaluation of blood flow velocity and flow direction can be carried out using Doppler sonography. Further evaluation of tumour perfusion can also be performed by low-mechanical contrast enhanced endoscopic ultrasound (CE-EUS). This is a high-resolution technique enabling minimally invasive evaluation of tumour perfusion.

According to the European Federation Societies in Ultrasound in Medicine and Biology (EFSUMB) guidelines, contrast enhanced-ultrasound (CE-EUS) can be utilized to assess early response to biologic therapy in tumours such as metastatic gastrointestinal stromal tumour (GIST) or renal cell carcinoma or hepatocellular carcinoma. A similar approach has not been tested yet in CRC patients using CE-EUS.

In this Ph.D. study the investigators have chosen to focus on left sided colonic cancers only, since they constitute approximately 70% of all colon cancers and, technically, are easier to reach than transverse tumours or right sided tumours, thereby making the study more feasible. The investigators have defined left sided colonic cancers as cancers including the left flexure proximally and until 15 cm from the linea Dentata distally.

Aims To examine if EUS can be used for stage assessment of left sided colon cancers and to investigate if endoscopic ultrasound perfusion assessment correlates to histopathological including immunohistochemical parameters of tumour vascular markers.

Project description The Ph.D. study consists of 4 sub-studies.

1. Endoscopic ultrasound for assessment of T-stage and N-stage in left-sided colonic cancers Hypothesis: EUS is a feasible staging method to accurately determine T-stage and N-stage in left-sided tumours.

   Objectives: To investigate left-sided colonic cancers with EUS especially concerning the muscular tumour invasion (tunica muscularis) and the detection rate of local lymph nodes suspicious of malignancy.

   Design: A prospective cohort study. Methods: Any patient at Køge/Roskilde and Herlev Hospital scheduled for surgery and with histologically determined left-sided colonic cancer will be included in the study and undergo EUS evaluation. Patients will undergo a CT-scan and will be staged preoperatively according to this scan. Sensitivity and specificity will be calculated for EUS and pathology specimens, regarding muscular invasion. It is expected, based on previous publications, that the distribution between patients with "bad" tumours (= T4 + T3 with > 5 mm muscular invasion) and "good" tumours (= T1 - T3 with < 5 mm muscular invasion) will be 45% and 55% respectively. With an 80% power and 5% type 1 error the investigators will include 74 patients in order to have an expected sensitivity of 90% and a lower boundary of the 95% confidence interval at 75%. The investigators will perform an interim analysis after inclusion of 35 patients. If the observed sensitivity will be below 80% the study will be terminated and there will be focus on method development. If the sensitivity will be higher than 80% the study inclusion will continue until inclusion of 74 patients.

   Outcome: Outcome measures will be EUS stage compared to histological stage as well as to CT scan stage.
2. The correlation between endoscopic perfusion assessments with immunohistochemical parameters in left sided colonic cancer Hypothesis: EUS is a feasible diagnostic modality to determine the vascular characteristics of left sided colonic cancer.

Objectives: To investigate quantitative and qualitative EUS parameters of left-sided colonic cancers with contrast enhanced EUS imaging.

Design: A prospective cohort study. Methods: When EUS staging has been performed in the cohort of study 2, further evaluation of tumour perfusion will be done by low-mechanical contrast enhanced endoscopic ultrasound (CE-EUS). Power Doppler vascularity index will be calculated and used as a measure of tumour perfusion. The volume of tumour perfusion has previously shown a strong correlation with the vascular density. The perfusion of tumour tissue per cm3 (automated pixel analysis) will be compared with histologically determined vascular density. The study is explorative and no sample size calculation is possible based on present literature.

Outcome: Outcome measures will be endoscopic ultrasound perfusion parameters correlated to histopathological vascular characteristics of left-sided colonic cancers (e.g. micro vessel density measured by CD31 staining and double-staining techniques).

Risks and side effects:

Complications may occur during EUS but they are rare. These consist of bleeding from the tumour, since tumour masses may be very vulnerable, when positioning the scope. The bleeding is self-limited. Perforation of the bowel is extremely rare. Making the EUS staging procedure and the endoscopic perfusion assessment will, all in all, take about 10-15 minutes. SonoVue® is not nephrotoxic and the incidence of hypersensitivity or severe allergic events is lower than with current X-ray agents and comparable to that of other magnetic resonance contrast agents. SonoVue® is approved for clinical use in EU countries and administration of the contrast agent showed very low incidence of side effects.

Location:

The data collection will take place at Department of Surgery, Endoscopy Units at Herlev University Hospital and Køge/Roskilde University Hospital. The endoscopies will be performed primarily at Herlev Hospital but also at Køge Hospital if necessary EUS equipment can be provided. If not patients from Køge and Roskilde Hospital will be examined at Herlev Hospital. The histopathological analyses follow the standard protocols for colorectal carcinomas routinely performed in the Departments of Pathology at Herlev University Hospital and Roskilde University Hospital.

Dissemination of the results:

All results, both positive, negative and inconclusive will be presented on national and international conferences. The results will be submitted for publication to peer-reviewed journals with Marie Louise Malmstrøm as the first author.

Sponsors:

The research project is initiated by the principal supervisor, Peter Vilmann, MD, DMSc. The costs associated with the project will be supported from the principal supervisor's department budget and external funding. The EUS equipment is already available at the endoscopy department of Herlev and funding for equipment for Køge/Roskilde Hospital have been applied for at the Research Council of the Region of Zealand. Funding for salary for the clinical investigator has been applied at private funds and public funds.

Ethics:

The study is ethically approved (H-4-2014-075) and approved at datatilsynet. The studies performed are registered in www.clinicaltrials.gov as requested by ICMJE (International Committee of Medical Journal Editors). Research subjects will have to give informed consent, based on written and oral information before inclusion in the study. Participants will be informed about any side-effects, risks or unplanned events that might occur during the implementation of the study. The minimal risks will be outweighed by the potential implications for future patient care. The study will be carried out with respect to the mental and physical integrity of the participants.

Guidelines in obtaining informed consent from participants:

Well informed signed consent from the research subjects is an essential criterion for inclusion in the trial. Both written and oral information will be provided to each candidate to the study by either the chief investigator or other health care persons that are qualified in explaining the project in detail. The patient will be made aware of the possibility of a second person (e.g. caregiver, relative) to be present at the interview. The interview will take place in a private room in order to provide an uninterrupted communication. At the interview the detailed information on the project will be covered, in oral and written form, including an easy-to-read presentation of the project with its predictable risks and side-effects, expected outcomes and benefits for the research.

The subjects will be entitled to some reflection time before giving consent (24-48 hours), taking care that the time limit stipulated for complete pretherapeutic evaluation of the cancer patient is not exceeded, and taking care that the project will not interfere with the routine clinical investigations and treatments of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for elective left-sided colon cancer surgery
* Age 18 to 100 years old, men or women
* Signed informed consent for EUS with contrast-enhancement

Exclusion Criteria:

* Prior treatment with chemo-radiotherapy (before the diagnosis of colon cancer)
* Prior endoscopic resection or attempted endoscopic resection (before the diagnosis of colon cancer, but in the same area as the cancer)
* Pregnant women
* Failure to provide informed consent
* Severe coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
T-stage in left sided colonic cancer determined by endoscopic ultrasound compared to histological stage | EUS examination, 10 min
  EUS stage compared to histological stage and CT scan stage

SECONDARY OUTCOMES:
Perfusion in left sided colonic cancer determined by contrast enhanced endoscopic ultrasound compared to histological vascular immunostaining | CE-EUS examination, 5 min
  Endoscopic ultrasound perfusion parameters correlated to histopathological vascular characteristics of left-sided colonic cancers

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vilmann, MD, DMSc, Study Director — Herlev Hospital
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev
  - Roskilde Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Unable to connect to PubMed to validate , last attempt on November 19, 2014 at 10:31 AM EST
- [Derived] Malmstrom ML, Saftoiu A, Riis LB, Hassan H, Klausen TW, Rahbek MS, Gogenur I, Vilmann P. Dynamic contrast-enhanced EUS for quantification of tumor perfusion in colonic cancer: a prospective cohort study. Gastrointest Endosc. 2018 Jun;87(6):1530-1538. doi: 10.1016/j.gie.2018.01.001. Epub 2018 Jan 9. PMID 29329991
- [Derived] Malmstrom ML, Gogenur I, Riis LB, Hassan H, Klausen TW, Perner T, Saftoiu A, Vilmann P. Endoscopic ultrasonography and computed tomography scanning for preoperative staging of colonic cancer. Int J Colorectal Dis. 2017 Jun;32(6):813-820. doi: 10.1007/s00384-017-2820-x. Epub 2017 Apr 21. PMID 28432444